CLINICAL TRIAL: NCT06634173
Title: The Diagnostic Value of FAPI PET/CT in Staging of Newly Diagnosed Prostate Cancer
Acronym: proFAPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M22PFI
Record Dates: First submitted 2023-09-20; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an interventional study without concurrent controls.
Masking Description: All scans will be reviewed by two senior nuclear medicine physicians (NWZ-Alkmaar and/or NCI-AVL), separately and blinded to any clinical information. If a consensus is not reached, a third observer is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FAPI PET/CT (Experimental): Patients will undergo an additional diagnostic FAPI PET/CT scan within four weeks after PSMA PET/CT and within four weeks before planned treatment.
  Interventions: Diagnostic Test: FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: FAPI PET/CT — This study applies the radiopharmaceutical 18Fluor-FAPI-74 (FAPI) for molecular imaging of FAP expression in vivo with FAPI PET/CT, to assess the presence and distribution of activated Cancer associated fibroblasts as a marker of Tumor Micro-Environment and indirectly as a marker for malignancies.
  Other Names: Fluor-18-FAPI-74

SUMMARY:
This study aims to investigate the diagnostic value of FAPI PET/CT, relative to standard-of-care imaging using PSMA PET/CT, in staging of newly diagnosed PCa. FAPI PET/CT will be visually and quantitatively correlated to PSMA PET/CT resulting in detection rates and target-to-background ratios. If available, histopathology of resected specimens will serve as reference test for operated patients in order to determine diagnostic accuracy. All outcomes are descriptive and serve as pilot for a potential subsequent larger prospective diagnostic study.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥ 18 years;
* WHO performance status 0, 1 or 2;
* Written informed consent;
* Biopsy-proven newly diagnosed PCa;
* International Society of Urological Pathology (ISUP) grade group (GG) ≥ 3 and/or PSA ≥ 20 ng/ml and/or ≥cT3a.

If all of the criteria above are met, a subject must also meet all of the following subgroup specific criteria:

Group 1 (n=15):

- PSMA PET/CT with PSMA-avid primary tumor with PSMA-avid loco-regional and/or distant metastases.

Group 2 (n=15):

* PSMA PET/CT with PSMA-avid primary tumor with no PSMA-avid loco-regional or distant metastases;
* Increased risk of nodal metastases according to the Briganti 2019 nomogram (Briganti ≥40%) [22];
* Scheduled for (laparoscopic) prostatectomy including ePLND.

Exclusion Criteria:

* Known second malignant disease that may complicate image interpretation.
* Inability to cooperate with the scan process: inability to lie relatively still and in supine for 30-60 minutes or patient body habitus above scanner dimensions.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
detection rates and target-to-background ratios of FAPI PET/CT in patients with hormone-sensitive PCa. | within four weeks after PSMA PET/CT and within four weeks before planned treatment.

SECONDARY OUTCOMES:
Diagnostic value of FAPI PET/CT, relative to PSMA PET/CT, in staging of newly diagnosed PCa | within four weeks after PSMA PET/CT and within four weeks before planned treatment.
Correlate histopathological findings after robot-assisted radical prostatectomy (RARP) with extended pelvic lymph node dissection (ePLND) to FAPI PET/CT findings to determine its diagnostic accuracy for staging of newly diagnosed PCa. | within four weeks after PSMA PET/CT and within four weeks before planned treatment.
Correlate laboratory parameters (prostate specific antigen (PSA) levels) after treatment to FAPI PET/CT findings to determine its diagnostic accuracy. | within four weeks after PSMA PET/CT and within four weeks before planned treatment.
Obtain preliminary data on the FAP overexpression in primary prostate tumor and lymph node metastases by immunohistochemical staining. | within four weeks after PSMA PET/CT and within four weeks before planned treatment.
Correlate immunohistochemical staining with FAPI uptake measured on PET/CT | within four weeks after PSMA PET/CT and within four weeks before planned treatment.

OTHER OUTCOMES:
Obtain preliminary data on the size of FAPI PET/CT-detectable pelvic lymph nodes | within four weeks after PSMA PET/CT and within four weeks before planned treatment.
Correlate biopsy Gleason score to the SUVmax of primary lesions on FAPI PET/CT. | within four weeks after PSMA PET/CT and within four weeks before planned treatment.
Correlate FAPI PET/CT findings to radiological findings on biparametric MRI (radiological T stage and PI-RADS assessment category). | within four weeks after PSMA PET/CT and within four weeks before planned treatment.